CLINICAL TRIAL: NCT05912374
Title: Implementing Cognitive Dysfunction Accommodation Strategies Into a Biobehavioral Pre-Exposure Prophylaxis (PrEP) Focused HIV Prevention Intervention for People Who Inject Drugs
Brief Title: Adapting a Behavioral Intervention to Accommodate Cognitive Dysfunction in People Who Inject Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Michael Copenhaver, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H22-0033
Record Dates: First submitted 2023-06-01; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: randomized controlled pilot trial
Who Masked: Participant
Masking Description: single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm with standard intervention (Active Comparator): Participants will complete a 4-week CHRP-BB standard intervention
  Interventions: Behavioral: standard Community-Friendly Health Recovery Program- Biobehavioral (CHRP-BB)
- Experimental arm with enhanced intervention (Experimental): Participants will complete a 4-week CHRP-BB intervention enhanced with included cognitive dysfunction accommodation strategies.
  Interventions: Behavioral: enhanced Community-Friendly Health Recovery Program- Biobehavioral (CHRP-BB)

INTERVENTIONS:
Behavioral: standard Community-Friendly Health Recovery Program- Biobehavioral (CHRP-BB) — CHRP-BB is an evidence-informed behavioral intervention for HIV prevention among high-risk drug users in treatment on PrEP. CHRP-BB consists of 4 weekly 50- minute sessions.
  Arms: Control arm with standard intervention
Behavioral: enhanced Community-Friendly Health Recovery Program- Biobehavioral (CHRP-BB) — The enhanced version of CHRP-BB is an adapted behavioral intervention for HIV prevention among high-risk drug users in treatment on PrEP. This intervention consists of 4 weekly 50- minute sessions that include cognitive dysfunction accommodation strategies.
  Arms: Experimental arm with enhanced intervention

SUMMARY:
The goal of this pilot work was to determine if the cognitive dysfunction accommodation strategies help patients retain/utilize more HIV prevention information and increase PrEP adherence. Fifty people who inject drugs (PWID) were prescribed PrEP and randomized to one of two conditions, Twenty-five PWID participated in a standard HIV prevention session and 25 other PWID participated in a HIV prevention session with the included accommodation strategies. At recruitment participants were asked to provide self-report of the screening form and cognitive functioning. The intervention consisted of a total of 5 sessions: 1 meeting to gain baseline information of participants and 4 intervention sessions. Participants completed the consent form, demographics, skills assessment, drug use behavior assessment, and HIV risk behavior assessment at the pre-interview meeting. Participants completed PrEP uptake assessments and skills assessments immediately following the intervention to compare the pre/post results between the two groups. All participants also completed an acceptability rating to help researchers determine the acceptability of the accommodation strategies used, at the end of the 4th session. The objective was to determine if the proposed accommodation strategies are feasible and efficacious at improving HIV prevention outcomes, including knowledge and skills. Information gleaned from this process will be used to refine the intervention approach for future testing and implementation.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years or older
* reported injection drug use in the past 30 days
* reported engagement in drug- and/or sex- related HIV risk behaviors
* HIV negative
* are willing to initiate PrEP use
* can communicate (read, write and speak) in English
* experience mild/moderate level of cognitive dysfunction

Exclusion Criteria:

* cannot attend all study sessions
* actively homicidal and/or suicidal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
HIV risk reduction skills assessment at baseline | pre intervention (week 0)
  a 15 item checklist of HIV risk reduction skills, the lower the score the lower the ability to perform HIV risk reduction skills
HIV risk reduction skills assessment, post intervention | post intervention (week 4)
  a 15 item checklist of HIV risk reduction skills, the lower the score the lower the ability to perform HIV risk reduction skills
number of participants who picked up PrEP prescription | post intervention (week 4)
  PrEP prescription filled by pharmacy

SECONDARY OUTCOMES:
number of participants recruited | pre intervention (week 0)
  Feasibility was measured via recruitment success
number of participants retained throughout study | post intervention (week 4)
  Feasibility was measured via retention success
Intervention Acceptability | post intervention (week 4)
  Participants completed an ten-item intervention acceptability rating, the lower the number the lower the participants acceptability of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Copenhaver, PhD, Principal Investigator — University of Connecticut
Locations (1):
- APT Foundation, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Mistler CB, Shrestha R, Copenhaver MM. Testing the feasibility, acceptability, and preliminary efficacy of integrating accommodation strategies into an HIV prevention intervention for people who inject drugs with cognitive dysfunction. J Subst Use Addict Treat. 2025 Feb;169:209582. doi: 10.1016/j.josat.2024.209582. Epub 2024 Nov 17. PMID 39551147